CLINICAL TRIAL: NCT05318976
Title: A Randomized, Placebo-Controlled, Double-Blind Study of XPro1595 in Patients With Early Alzheimer's Disease With Biomarkers of Inflammation
Brief Title: A Study of XPro1595 in Patients With Early Alzheimer's Disease With Biomarkers of Inflammation
Acronym: MINDFuL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPro1595-AD-02
Record Dates: First submitted 2022-03-07; First posted 2022-04-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Mild Cognitive Impairment
Keywords: Inflammation; Biomarker; TNF
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Cognitive Dysfunction; Inflammation | interventions — XENP 1595

STUDY DESIGN:
Intervention Model Description: * (2:1) XPro1595 (1mg/kg), placebo
  * Weekly subcutaneous injections
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.0 mg/kg XPro1595 (Experimental): 1.0 mg/kg of XPro1595 will be administered via subcutaneous injection once a week for 23 weeks.
  Interventions: Drug: XPro1595
- 1.0 mg/kg Placebo (Placebo Comparator): 1.0 mg/kg of Placebo will be administered via subcutaneous injection once a week for 23 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XPro1595 — XPro1595 will be delivered by subcutaneous injection once a week
  Other Names: INB03/XPro™; XENP1595; DN-TNF
  Arms: 1.0 mg/kg XPro1595
Drug: Placebo — Placebo will be delivered by subcutaneous injection once a week
  Other Names: Matching Placebo
  Arms: 1.0 mg/kg Placebo

SUMMARY:
The goal of this Phase 2 Alzheimer's study is to determine whether 1.0 mg/kg XPro1595 confers a benefit on cognition, function, and biomarkers of white matter and to further evaluate safety and tolerability. The objectives of this study are to determine the safety, tolerability, and efficacy of XPro1595 in patients with early ADi.

DETAILED DESCRIPTION:
This trial is a randomized clinical study using XPro1595 to treat patients with Early Alzheimer's Disease with biomarkers of inflammation (ADi). Early ADi patients are defined as patients with Mild Alzheimer's Disease or Mild Cognitive Impairment (MCI) with a biomarker of inflammation.

ELIGIBILITY:
The screening window for this trial is 45 days.

Inclusion Criteria:

To be eligible for study entry, patients must satisfy all of the following criteria:

* Adult patients 50 years to ≤ 85 years of age at the time of consent;
* Meets the diagnostic criteria of MCI of probable Alzheimer's disease (Jack et al. 2018; NIA-AA) or mild dementia as clinically described in McKhann, (2011) and corresponding to stages 3 or 4 of the revised AD staging system (Jack, 2018). (NIA-AA);
* Amyloid positive (documented in medical history or assessed during screening through blood test);
* Either currently or previously (in pre-AD condition) literate and capable of reading, writing, and communicating effectively with others;
* Residence in an assisted living is allowed as is personal assistances provided in the home, however at time of enrollment participant must be able to perform most ADL with minimal assistance, and participant must be permitted sufficient independence to allow assessment of change in ADL;
* Has a study partner for the duration of the trial who either lives in the same household or interacts with the patient at least 4 hours per day and on at least 4 days per week, who is knowledgeable about the patient's daytime and night-time behaviors and who can be available to attend all clinic visits in person at which caregiver assessments are performed.

Exclusion Criteria:

Patients will be excluded from the study if 1 or more of the following criteria are applicable:

* Have any contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (e.g., in-skull and cardiac devices other than those approved as safe for use in MRI scanners);
* Receives considerable help to carry out basic ADL living either in the home or as a resident in a nursing home or similar facility;
* Lifetime history of a major psychiatric disorder including schizophrenia and bipolar disorder. Major depressive disorder that has resulted in 2 or more hospitalizations in a lifetime. Major depressive episode during the past 5 years that is judged by the clinical team unlikely to have been part of Alzheimer's prodrome. History of suicidality.
* History of substance abuse within 12 months; use of cannabis or cannabis products within 6 months of consent;
* Enrolled in another clinical trial where patients receive treatment with an investigational drug or treatment device or have had previous treatment with any investigational medicinal product within 60 days or 5 half-lives (whichever is longer) prior to study drug treatment;
* A prior organ or stem cell transplant;
* Seated blood pressure of ≥ 165/105 mmHg at Screening.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Early and Mild Alzheimer's Cognitive Composite (EMACC) | 24 Weeks
  Change in the Early and Mild Alzheimer's cognitive composite (EMACC) from Baseline to Week 24 in the following assessments:
  * International Shopping List Test-Immediate recall (Word List learning Test)
  * Digit Span Forward and Backward
  * Category Fluency Test (DKEFS)
  * Letter Fluency Test (DKEFS)
  * Trail Making Test Parts A and B
  * Digit Symbol Coding Test
  To assess the efficacy of XPro1595 compared with placebo on cognitive performance in patients with early ADi

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating (CDR) | 24 Weeks
  Change from Baseline to Week 24 in Clinical Dementia Rating Scale (CDR)
  The CDR scale is a clinician-rated dementia staging system that tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgement, and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5-point scale in which None = 0, Questionable = 0.5, Mild = 1, Moderate = 2, and Severe = 3. The global CDR score is established by clinical scoring rules and has values of 0 (no dementia), 0.5, (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). The Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment.
  To assess the effect of XPro1595 compared with placebo on cognition and global function in patients with early ADi
Change in apparent fiber density (AFD) | 24 Weeks
  Change from Baseline to Week 24 in apparent fiber density (AFD)
  To assess the efficacy of XPro1595 compared with placebo on axonal integrity in patients with early ADi
Change in Everyday Cognition (E-Cog) | 24 Weeks
  Change from Baseline to Week 24 in Everyday Cognition (E-Cog)
  To evaluate the effect of XPro1595 compared with placebo on E-Cog
Change in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-MCI-ADL) | 24 Weeks
  Change from Baseline to Week 24 in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-MCI-ADL)
  To assess the effect of XPro1595 compared with placebo on ADL in patients with early ADi.
Change in myelin content | 24 Weeks
  Change from Baseline to Week 24 in free-water-corrected tissue Radial diffusivity and 1 of the following i) MRI-specific myelin contrast: ii) a magnetization transfer ratio (MTR) iii) an inhomogeneous magnetization transfer (MT) or iv) an myelin water fraction (MWF) map
  To assess the efficacy of XPro1595 compared with placebo on myelin in patients with early ADi.
Change in non-cognitive behavioral symptoms | 24 Weeks
  Change from Baseline to Week 24 in (Neuropsychiatric Inventory [NPI] caregiver items)
  To assess the effect of XPro1595 compared with placebo on noncognitive behavioral symptoms in patients with early ADi
Change in gray matter integrity | 24 Weeks
  Change from Baseline to Week 24 in Cortical Disarray Measurement (CDM®)
  To assess the efficacy of XPro1595 compared with placebo on gray matter integrity in patients with early ADi
Change in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid) | 24 Weeks
  Number of participants with a reduction in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration amyloid) from Baseline to Week 24.
  To assess the efficacy of XPro1595 compared with placebo on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid).
Change in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau) | 24 Weeks
  Change from Baseline to Week 24 in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau)
  To assess the efficacy of XPro1595 compared with placebo on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau)
Change in brain structure neurodegeneration | 24 Weeks
  Changes from Baseline to Week 24 in volumetric magnetic resonance imaging (MRI)
  To assess the efficacy of XPro1595 compared with placebo on brain structure neurodegeneration
Number of participants who experience adverse events and serious adverse events | Baseline up to 28 days post last dose
  Clinically significant abnormalities of laboratory values, physical findings, electrocardiogram findings and other safety assessments will be recorded as adverse events if the findings meet the defined criteria for adverse events.

OTHER OUTCOMES:
Change in Goal Attainment Scale (GAS) | 24 Weeks
  Change in individual goals based on the Goal Attainment Scale (GAS)
  The achievement of each goal is rated on a 5-point attainment scale (-2, -1, 0, +1, +2) to allow standardized scoring of personalized outcomes. A participant's overall goal attainment is quantified using a formula that takes into account the number of goals that have been set, and the extent to which they are correlated with each other. For each identified goal area, the caregiver will be asked to give a detailed description of the patient's current (baseline) status and goal status, which will be recorded at the -1 and 0 levels on the 5-point scale, respectively. The remaining levels of the scale will then be set: somewhat better than the goal (+1), much better than the goal (+2), and much worse than the goal (-2).
  To evaluate the effect of XPro1595 compared with placebo on goal attainment scores

CONTACTS AND LOCATIONS:
Overall Officials: Therese Blomberg, Study Director — INmune Bio
Locations (37):
- Australia (8):
  - INmune Bio Investigational Site, Darlinghurst, New South Wales
  - INmune Bio Investigational Site, Macquarie Park, New South Wales
  - INmune Bio Investigational Site, Adelaide, South Australia
  - INmune Bio Investigational Site, Box Hill, Victoria
  - INmune Bio Investigational Site, Carlton, Victoria
  - INmune Bio Investigational Site, Ivanhoe, Victoria
  - INmune Bio Investigational Site, Parkville, Victoria
  - INmune Bio Investigational Site, Nedlands, Western Australia
- Canada (5):
  - INmune Bio Investigational Site, Kelowna
  - INmune Bio Investigational Site, Ottawa
  - INmune Bio Investigational Site, Sherbrooke
  - INmune Bio Investigational Site, Toronto
  - INmune Bio Investigational Site, West Vancouver
- Czechia (4):
  - INmune Bio Investigational Site, Brno
  - INmune Bio Investigational Site, Pilsen
  - INmune Bio Investigational Site, Prague
  - INmune Bio Investigational Site, Rychnov nad Kněžnou
- France (3):
  - INmune Bio Investigational Site, Bron
  - INmune Bio Investigational Site, Nantes
  - INmune Bio Investigational Site, Toulouse
- Germany (2):
  - INmune Bio Investigational Site, Berlin
  - INmune Bio Investigational Site, Chemnitz
- Poland (3):
  - INmune Bio Investigational Site, Bialystok
  - INmune Bio Investigational Site, Bydgoszcz
  - INmune Bio Investigational Site, Wroclaw
- Spain (5):
  - INmune Bio Investigational Site, Barcelona
  - INmune Bio Investigational Site, Córdoba
  - INmune Bio Investigational Site, Madrid
  - INmune Bio Investigational Site, Seville
  - INmune Bio Investigational Site, Valencia
- United Kingdom (7):
  - INmune Bio Investigational Site, Birmingham
  - INmune Bio Investigational Site, Bristol
  - INmune Bio Investigational Site, Guildford
  - INmune Bio Investigational Site, London
  - INmune Bio Investigational Site, Motherwell
  - INmune Bio Investigational Site, Plymouth
  - INmune Bio Investigational Site, Winchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bongartz T, Sutton AJ, Sweeting MJ, Buchan I, Matteson EL, Montori V. Anti-TNF antibody therapy in rheumatoid arthritis and the risk of serious infections and malignancies: systematic review and meta-analysis of rare harmful effects in randomized controlled trials. JAMA. 2006 May 17;295(19):2275-85. doi: 10.1001/jama.295.19.2275. PMID 16705109
- [Background] Chance SA, Clover L, Cousijn H, Currah L, Pettingill R, Esiri MM. Microanatomical correlates of cognitive ability and decline: normal ageing, MCI, and Alzheimer's disease. Cereb Cortex. 2011 Aug;21(8):1870-8. doi: 10.1093/cercor/bhq264. Epub 2011 Jan 14. PMID 21239393
- [Background] Chou RC, Kane M, Ghimire S, Gautam S, Gui J. Treatment for Rheumatoid Arthritis and Risk of Alzheimer's Disease: A Nested Case-Control Analysis. CNS Drugs. 2016 Nov;30(11):1111-1120. doi: 10.1007/s40263-016-0374-z. PMID 27470609
- [Background] Clark I, Atwood C, Bowen R, Paz-Filho G, Vissel B. Tumor necrosis factor-induced cerebral insulin resistance in Alzheimer's disease links numerous treatment rationales. Pharmacol Rev. 2012 Oct;64(4):1004-26. doi: 10.1124/pr.112.005850. Epub 2012 Sep 10. PMID 22966039
- See also: Alzheimer's Association annual report releasing statistics regarding Alzheimer's disease — https://www.alz.org/alzheimers-dementia/facts-figures